CLINICAL TRIAL: NCT01068054
Title: A Double-blind Comparison of 0.1% Tacrolimus Ophthalmic Ointment and 2% Cyclosporine Eye Drops in the Treatment of Vernal Keratoconjunctivits (VKC)
Brief Title: Efficacy Study of FK-506 and Cyclosporine in Vernal Keratoconjunctivits (VKC)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Pakit Vichyanond, MD, Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: fk506vscyclosporine_vkc
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2003-06

CONDITIONS: Keratoconjunctivitis, Vernal
Keywords: vernal keratoconjunctivitis; FK-506; tacrolimus; cyclosporine; children
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Tacrolimus; Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tacrolimus (Active Comparator): Tacrolimus arm: active 0.1% tacrolimus eye ointment BID + placebo eye drops QID
  Interventions: Drug: tacrolimus
- cyclosporine (Active Comparator): 2% cyclosporine eye drops apply QID + placebo eye ointment apply bid
  Interventions: Drug: cyclosporins

INTERVENTIONS:
Drug: tacrolimus — 0.1% ointment,apply bid, 8 weeks
  Arms: tacrolimus
Drug: cyclosporins — 2% eyclosporine eye drops apply 1 drop to each eye QID
  Arms: cyclosporine

SUMMARY:
The study was a double-blind, parallel study to compare efficacy of 0.1% tacrolimus ophthalmic ointment vs 2% cyclosporine eye drops in children with vernal keratoconjunctivitis. The duration of the blinded period was 8 weeks followed with 4 weeks of open-period of tacrolimus ointment. The hypothesis was that tacrolimus was as effective as cyclosporine for the treatment of this condition.

DETAILED DESCRIPTION:
Background: Vernal keratoconjunctivitis (VKC) is a serious, sight-threatening ocular disease, occurring mainly in children. Prolonged use of ophthalmic corticosteroids is usually required in severe cases which could lead to serious complications such as glaucoma and cataract. Cyclosporine and tacrolimus are among newer treatments for VKC.

Objective: To compare the efficacy of 0.1% tacrolimus (FK-506) ophthalmic ointment with 2% cyclosporine eye drops in the treatment of VKC.

Methods: Twenty-four patients with VKC were recruited. After a 2 week-washout period, they were randomized into 2 groups in a double-blinded, parallel fashion. The first group received 0.1% FK-506 eye ointment with placebo eye drops and the second group received 2% cyclosporine eye drops with placebo ointment for 8 weeks. Thereafter, all patients received an open-treatment with 0.1% FK-506 eye ointment for another 4 weeks. Subjective ocular symptoms and side effects were scored by patients at the entry, and at the end of the 1st, 4th, 8th and 12th weeks. Objective ocular signs were evaluated by an ophthalmologist (PK) at all follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinical diagnosis of vernal keratoconjunctivitis

Exclusion Criteria:

* coexisting ocular diseases such as glaucoma, other corneal disease, ocular infections, other coexisting systemic diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-06; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
overall subjective ocular symptom scores | 8 weeks

SECONDARY OUTCOMES:
overall objective ocular signs | 8 weeks
overall side-effect scores | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pakit Vichyanond, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Bangkok, Thailand